CLINICAL TRIAL: NCT01714622
Title: Prospective Cohort Study for Analyzing the Effect of Gastric Cancer Surgery to the Metabolic Syndrome and Insulin Resistance
Status: Withdrawn | Type: Observational
Why Stopped: Canceled study due to delay of progress procedure and failure to obtain research funds.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0550
Record Dates: First submitted 2012-10-17; First posted 2012-10-26 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2015-09

CONDITIONS: Gastric Cancer With Metabolic Syndrome or Metabolic Disease
Keywords: metabolic syndrome; insulin resistance; gastric cancer
MeSH Terms: conditions — Metabolic Diseases; Metabolic Syndrome; Insulin Resistance; Stomach Neoplasms | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- metabolic syndrome: gastric cancer patients with metabolic syndrome
  Interventions: Procedure: subtotal gastrectomy with gastroduodenostomy; Procedure: subtotal gastrectomy with Roux-en-Y gastrojejunostomy,; Procedure: total gastrectomy with Rou-en-Y esophagojejunostomy
- metabolic disease: gastric cancer patients with metabolic disease
  Interventions: Procedure: subtotal gastrectomy with gastroduodenostomy; Procedure: subtotal gastrectomy with Roux-en-Y gastrojejunostomy,; Procedure: total gastrectomy with Rou-en-Y esophagojejunostomy
- normal: gastric cancer patients without metabolic syndrome or metabolic disease
  Interventions: Procedure: subtotal gastrectomy with gastroduodenostomy; Procedure: subtotal gastrectomy with Roux-en-Y gastrojejunostomy,; Procedure: total gastrectomy with Rou-en-Y esophagojejunostomy

INTERVENTIONS:
Procedure: subtotal gastrectomy with gastroduodenostomy
Procedure: subtotal gastrectomy with Roux-en-Y gastrojejunostomy,
Procedure: total gastrectomy with Rou-en-Y esophagojejunostomy

SUMMARY:
Gastric cancer is still one of the most common malignance in Korea. Because of the popularity of regular check ups, early detection of gastric cancer has increased, consequently, the survival of the patients also has increased. In this reason, the interest of outcomes after gastrectomy for gastric cancer move survival only to quality of life of these patients.

Although the definition of metabolic syndrome is various, but it is normally accepted as a state that insulin resistance or glucose intolerance combined with hypertension or hyperlipidemia or obesity. Metabolic syndrome is a worldwide health problem, and the treatment is modification of life style, weight loss and medication. However, in most of the patients metabolic syndrome is considered not curable disease. Recent studies have shown that some bariatric surgery offers not only control the overweight but also metabolic syndrome. The exact mechanism is still unknown but decreased gastric volume and intestinal bypass itself seemed to play an important role to improve metabolic syndrome over just decreased weight.

For treating gastric cancer, gastrectomy is essential and the extent of gastrectomy is varied subtotal and total gastrectomy according to the location of tumor. Also, reconstruction type is varied gastroduodenostomy and Roux-en-Y gastrojejunostomy after subtotal gastrectomy, esophagojejunostomy after total gastrectomy. This kind of operation for gastric cancer lead decreased gastric volume and/or intestinal bypass, which means this operation could lead similar effect of bariatric surgery. Already, there have been several retrospective reports that metabolic syndrome or diabetes was improved after gastrectomy for gastric cancer but no prospective study about this subject yet in Korea.

The purpose of this study is that evaluating the degree of improvement of metabolic syndrome after gastrectomy for gastric cancer, and analyze the differences between the type of operation.

ELIGIBILITY:
Inclusion Criteria:

1. gastric cancer,
2. in plan for gastrectomy for gastric cancer
3. ages between 20 to 85 years old
4. assign in consent

Exclusion Criteria:

1. vulnerable subject (pregnant, be devoid of mental capacity, soldiers, or medical students)
2. had low performance scale due to severe cardiovascular disease.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: in plan to underwent curative gastrectomy for gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
the changes of metabolic syndrome | baseline to postoperative 3 month, and there after every 6 months until 24 months after the gastrectomy

SECONDARY OUTCOMES:
the changes of insulin resistance after gastrectomy | baseline to postoperative 3 month, and there after every 6 months until 24 months after the gastrectomy

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Department of Surgery, Yonsei University Colleage of Medicine,, Seoul
  - Ji Yeong An, Seoul
  - Sevrance hospital, Department of General surgery, Seoul